CLINICAL TRIAL: NCT02468674
Title: A 24 Week Off Drug Extension, Parallel Group, Study Assessing Durability of Effect on Skeletal Muscle Strength and Function Following a 6-month Double-blind, Placebo Controlled Study Evaluating Bimagrumab in Older Adults With Sarcopenia (InvestiGAIT Extension)
Brief Title: A 24-week Off-drug Extension Study in Sarcopenic Elderly Who Completed Treatment in the 6-month Core Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYM338E2202E1; 2015-000471-27 (EudraCT Number)
Record Dates: First submitted 2015-04-30; First posted 2015-06-11 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Sarcopenia
Keywords: Sarcopenia, muscle wasting, elderly, strength, physical function, lean body mass, gait speed
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Follow-up (arm 1) (Other): Patients in Population I received 6 doses of bimagrumab 70 mg, 210 mg, 700 mg or placebo - one approximately every four weeks - over a 20-week period providing drug exposure for a total of 24 weeks.
  Interventions: Drug: bimagrumab; Drug: Placebo
- Follow-up (arm 2) (No Intervention): Patients in Population II received either bimagrumab 700 mg or placebo in the core study and did not receive any investigational treatment in the extension study.

INTERVENTIONS:
Drug: bimagrumab — bimagrumab low dose bimagrumab moderate dose bimagrumab high dose
  Patients enrolled prior to the protocol amendment 1 (Population I ), who received bimagrumab in the core study, entered the extension study at Week 25 and were randomly assigned to two subgroups within each of three treatment arms to either receive bimagrumab at the same dose level or placebo. Study medication was administered as an intravenous infusion starting at Week 25 after treatment was initiated in the core study until week 45.
  Arms: Follow-up (arm 1)
Drug: Placebo — Placebo
  Patients enrolled prior to the protocol amendment 1 (Population I), who received placebo in core study, entered the extension study at Week 25 and received placebo as an intravenous infusion starting at Week 25 after treatment was initiated in the core study until week 45.
  Arms: Follow-up (arm 1)

SUMMARY:
This extension study was a 24-week off-drug follow-up of the core CBYM338E2202 (NCT ) study and the main objective was to determine the long-term durability of bimagrumab (BYM338) effect after a 6-month treatment period.

DETAILED DESCRIPTION:
Two populations were defined as below:

* Population I: Patients enrolled prior to the protocol amendment 1, who received bimagrumab 70 mg, 210 mg or 700 mg in the core study, were randomly assigned to two subgroups within each of three treatment arms to either receive bimagrumab at the same dose level or placebo. Patients receiving placebo in the core study continued receiving placebo in the extension study.
* Population II: Patients enrolled after protocol amendment 1, who received bimagrumab 700 mg or placebo in the core study, did not receive study medication in the extension study and were followed-up per schedule defined in this protocol amendment.

ELIGIBILITY:
Inclusion criterion:

- Men and postmenopausal women aged 70 years or older that have participated in, and have completed the full study treatment period per protocol (24 weeks/EOT visit) in the preceding core study (CBYM338E2202)

Exclusion criterion:

- Any condition which should have led to treatment discontinuation per protocol in the core study (CBYM338E2202)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (5):
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Gainesville, Georgia
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, St Albans, Victoria, Australia
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Copenhagen NV, Denmark
- France (2):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Pessac
- Japan (10):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Nara, Nara
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Kitaadachigun Inamachi, Saitama
  - Novartis Investigative Site, Kitamoto, Saitama
  - Novartis Investigative Site, Itabashi Ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Koto-ku, Tokyo
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Suwon, Gyeonggi-do, South Korea
- Spain (2):
  - Novartis Investigative Site, Albacete, Castille-La Mancha
  - Novartis Investigative Site, Getafe, Madrid
- Novartis Investigative Site, Geneva, Switzerland
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 30 centers in 12 countries: Australia (1), Belgium (1), Czech Republic (1), Denmark (1), France (2), Japan (10), Russia (4), South Korea (1), Spain (2), Switzerland (1), Taiwan (1), United States (5).
Groups:
- Population I: BYM338 700 mg; Population I BYM338: 700 mg to Placebo; Population I: BYM338 210 mg; Population I BYM338: 210 mg to Placebo; Population I: BYM338 70 mg; Population I: BYM338 70 mg to Placebo; Population I: Placebo: Follow-up (arm 1): Patients in Population I received 6 doses of bimagrumab 70 mg, 210 mg, 700 mg or placebo - one approximately every four weeks - over a 20-week period providing drug exposure for a total of 24 weeks.
- Population: II BYM338 700 mg; Population: II Placebo: Follow-up (arm 2): Patients in Population II received either bimagrumab 700 mg or placebo in the core study and did not receive any investigational treatment in the extension study.
Period: Overall Study
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo | Population: II BYM338 700 mg | Population: II Placebo
Started (All randomized patients were included in the Full Analysis (FAS) and Safety Set) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 69 | 43
Completed | 4 | 5 | 5 | 3 | 6 | 6 | 14 | 65 | 40
Not Completed | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient/Guardian Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
Groups:
- Total: Total of all reporting groups
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo | Population: II BYM338 700 mg | Population: II Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 69 | 43 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age Continuous for Population I Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Years
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    (all) | 80.0 (4.90) | 79.4 (7.27) | 79.0 (1.58) | 74.8 (2.63) | 77.6 (6.75) | 81.6 (4.58) | 79.9 (4.22) |  |  | 79.2 (4.91)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age Continuous for Population II Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    (all) |  |  |  |  |  |  |  | 79.8 (5.05) | 78.2 (5.29) | 79.2 (5.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender for Population I Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    Female | 1 | 2 | 2 | 2 | 3 | 5 | 8 | 0 | 0 | 23
    Male | 4 | 3 | 3 | 2 | 4 | 2 | 7 | 0 | 0 | 25
Sex: Female, Male [Count of Participants; unit: Participants] — Gender for Population II Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 29 | 69
    Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 14 | 43
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity for Population I Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Participants
    Asian: number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    Asian | 1 | 0 | 0 | 1 | 2 | 2 | 6 |  |  | 12
    Black: number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    Black | 0 | 0 | 0 | 0 | 1 | 1 | 1 |  |  | 3
    Caucasian: number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    Caucasian | 4 | 5 | 5 | 3 | 4 | 4 | 8 |  |  | 33
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity for Population II Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Participants
    Asian: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    Asian |  |  |  |  |  |  |  | 11 | 3 | 14
    Caucasian: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    Caucasian |  |  |  |  |  |  |  | 56 | 40 | 96
    Native American: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    Native American |  |  |  |  |  |  |  | 1 | 0 | 1
    Pacific Islander: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    Pacific Islander |  |  |  |  |  |  |  | 1 | 0 | 1
Population I: Short Physical Performance Battery (SPPB) total score at Week 25 [Mean (Standard Deviation); unit: Scores on a scale] — Baseline Extension Visit = Week 25. SPPB evaluates lower extremities in three functional components: maintenance of standing balance, usual gait speed and chair stand. Each test yields a score on a scale from 0 to 4 (total score 0-12, with the higher score reflecting a higher level of function). Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Scores on a scale
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    (all) | 8.8 (2.17) | 10.4 (1.34) | 8.6 (1.67) | 8.5 (1.91) | 8.9 (2.04) | 8.0 (3.27) | 9.1 (1.58) |  |  | 8.9 (2.01)
Population II: Short Physical Performance Battery (SPPB) total score at Week 25 [Mean (Standard Deviation); unit: Scores on a scale] — Baseline Extension Visit = Week 25. SPPB evaluates lower extremities in three functional components: maintenance of standing balance, usual gait speed and chair stand. Each test yields a score on a scale from 0 to 4 (total score 0-12, with the higher score reflecting a higher level of function). Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  Scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    (all) |  |  |  |  |  |  |  | 8.5 (2.17) | 8.2 (2.25) | 8.4 (2.20)
Population I: 6-minute walking distance (6MWT) at Week 25 [Mean (Standard Deviation); unit: meters] — Baseline Extension Visit = Week 25. The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway. Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  meters
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    (all) | 302.73 (130.22) | 353.10 (66.17) | 313.67 (71.39) | 361.07 (80.11) | 305.24 (111.34) | 286.94 (119.37) | 352.18 (123.55) |  |  | 327.49 (106.64)
Population II: 6-minute walking distance (6MWT) at Week 25 [Mean (Standard Deviation); unit: meters] — Baseline Extension Visit = Week 25. The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway. Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  meters
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    (all) |  |  |  |  |  |  |  | 307.84 (99.96) | 315.61 (95.74) | 310.81 (98.01)
Population I: Gait speed at Week 25 [Mean (Standard Deviation); unit: m/sec] — Baseline Extension Visit = Week 25. Gait Speed was assessed as part of SPPB, over a 4 meter distance of a 6 meter course. Gait speed assesses a person's usual walking speed, which is defined as the speed a person normally walks from one place to another. Poor functional performance is measured by slow or declining gait speed. Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  m/sec
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15 | 0 | 0 | 48
    (all) | 0.8 (0.20) | 0.9 (0.13) | 0.9 (0.27) | 0.9 (0.12) | 0.8 (0.19) | 0.6 (0.28) | 0.8 (0.19) |  |  | 0.8 (0.21)
Population II: Gait speed at Week 25 [Mean (Standard Deviation); unit: m/sec] — Baseline Extension Visit = Week 25. Gait Speed was assessed as part of SPPB, over a 4 meter distance of a 6 meter course. Gait speed assesses a person's usual walking speed, which is defined as the speed a person normally walks from one place to another. Poor functional performance is measured by slow or declining gait speed. Population: 160 participants were enrolled into the study: 48 in Population I (patients enrolled prior to protocol amendment 1) and 112 in Population II (patients enrolled after protocol amendment 1)
  m/sec
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 43 | 112
    (all) |  |  |  |  |  |  |  | 0.8 (0.23) | 0.8 (0.22) | 0.8 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Population I: Short Physical Performance Battery (SPPB) Total Score at Week 49
Description: SPPB evaluates lower extremities in three functional components: maintenance of standing balance, usual gait speed and chair stand. Each test yields a score on a scale from 0 to 4 (total score 0-12, with the higher score reflecting a higher level of function).
Time Frame: Week 49
Population: The Full Analysis Set (FAS), which consisted of all randomized patients to whom study treatment had been assigned, was considered. For post Week 25 assessments, only the subjects with assessment available at both the Visit and Week 25 are included in the calculation of the respective Visit statistics.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo
Number analyzed (Participants) | 4 | 5 | 5 | 3 | 6 | 6 | 14
Scores on a scale | 8.8 (3.86) | 10.2 (1.92) | 8.0 (2.35) | 8.0 (2.65) | 9.5 (2.17) | 7.5 (3.78) | 9.6 (1.83)
Statistical Analysis 1: Comparison: Population I: BYM338 700 mg vs Population I BYM338: 700 mg to Placebo; Population I: SPPB total score at Week 49; Test type: Other; p = 0.759, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 2: Comparison: Population I: BYM338 210 mg vs Population I BYM338: 210 mg to Placebo; Population I: SPPB total score at Week 49; Test type: Other; p = 0.500, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 3: Comparison: Population I: BYM338 70 mg vs Population I: BYM338 70 mg to Placebo; Population I: SPPB total score at Week 49; Test type: Other; p = 0.144, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 4: Comparison: Population I: BYM338 700 mg vs Population I: Placebo; Population I: SPPB total score at Week 49; Test type: Other; p = 0.648, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 5: Comparison: Population I: BYM338 210 mg vs Population I: Placebo; Population I: SPPB total score at Week 49; Test type: Other; p = 0.929, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 6: Comparison: Population I: BYM338 70 mg vs Population I: Placebo; Population I: SPPB total score at Week 49; Test type: Other; p = 0.530, t-test, 1 sided; One-sided test at the 0.025 significance

2. Primary Outcome: Population II: Short Physical Performance Battery (SPPB) Total Score at Week 49
Description: as for outcome 1
Time Frame: Week 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Population: II BYM338 700 mg | Population: II Placebo
Number analyzed (Participants) | 65 | 40
Scores on a scale | 8.6 (2.40) | 8.8 (1.55)
Statistical Analysis 1: Comparison: Population: II BYM338 700 mg vs Population: II Placebo; Population II: SPPB total score at Week 49; Test type: Other; p = 0.839, ANCOVA; Difference in the least square means (SE)

3. Secondary Outcome: Population I: 6-minute Walking Distance (6MWT) at Week 49
Description: The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway. A high 6MWT represent better physical condition.
Time Frame: Week 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15
meters | 318.2 (159.55) | 354.1 (69.98) | 304.1 (63.05) | 361.5 (144.53) | 316.1 (97.87) | 273.4 (154.03) | 368.7 (108.37)
Statistical Analysis 1: Comparison: Population I: BYM338 700 mg vs Population I BYM338: 700 mg to Placebo; Population I: 6MWT at Week 49; Test type: Other; p = 0.669, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 2: Comparison: Population I: BYM338 210 mg vs Population I BYM338: 210 mg to Placebo; Population I: 6MWT at Week 49; Test type: Other; p = 0.773, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 3: Comparison: Population I: BYM338 70 mg vs Population I: BYM338 70 mg to Placebo; Population I: 6MWT at Week 49; Test type: Other; p = 0.290, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 4: Comparison: Population I: BYM338 700 mg vs Population I: Placebo; Population I: 6MWT at Week 49; Test type: Other; p = 0.766, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 5: Comparison: Population I: BYM338 210 mg vs Population I: Placebo; Population I: 6MWT at Week 49; Test type: Other; p = 0.885, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 6: Comparison: Population I: BYM338 70 mg vs Population I: Placebo; Population I: 6MWT at Week 49; Test type: Other; p = 0.840, t-test, 1 sided; One-sided test at the 0.025 significance level

4. Secondary Outcome: Population II: 6-minute Walking Distance (6MWT) at Week 49
Description: as for outcome 3
Time Frame: Week 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Population: II BYM338 700 mg | Population: II Placebo
Number analyzed (Participants) | 69 | 43
meters | 321.2 (105.13) | 323.1 (96.47)
Statistical Analysis 1: Comparison: Population: II BYM338 700 mg vs Population: II Placebo; Population II: 6MWT at Week 49; Test type: Other; p = 0.367, ANCOVA; Difference in the least square means (SE)

5. Secondary Outcome: Population I: Gait Speed at Week 49
Description: Gait Speed was assessed as part of SPPB, over a 4 meter distance of a 6 meter course. Gait speed assesses a person's usual walking speed, which is defined as the speed a person normally walks from one place to another. Poor functional performance is measured by slow or declining gait speed.
Time Frame: Week 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15
m/sec | 0.8 (0.35) | 1.0 (0.18) | 0.9 (0.17) | 1.1 (0.24) | 0.9 (0.15) | 0.7 (0.35) | 0.8 (0.18)
Statistical Analysis 1: Comparison: Population I: BYM338 700 mg vs Population I BYM338: 700 mg to Placebo; Population I: Gait speed at Week 49; Test type: Other; p = 0.875, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 2: Comparison: Population I: BYM338 210 mg vs Population I BYM338: 210 mg to Placebo; Population I: Gait speed at Week 49; Test type: Other; p = 0.909, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 3: Comparison: Population I: BYM338 70 mg vs Population I: BYM338 70 mg to Placebo; Population I: Gait speed at Week 49; Test type: Other; p = 0.168, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 4: Comparison: Population I: BYM338 700 mg vs Population I: Placebo; Population I: Gait speed at Week 49; Test type: Other; p = 0.632, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 5: Comparison: Population I: BYM338 210 mg vs Population I: Placebo; Population I: Gait speed at Week 49; Test type: Other; p = 0.310, t-test, 1 sided; One-sided test at the 0.025 significance
Statistical Analysis 6: Comparison: Population I: BYM338 70 mg vs Population I: Placebo; Population I: Gait speed at Week 49; Test type: Other; p = 0.321, t-test, 1 sided; One-sided test at the 0.025 significance

6. Secondary Outcome: Population II: Gait Speed at Week 49
Description: as for outcome 5
Time Frame: Week 49
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Population: II BYM338 700 mg | Population: II Placebo
Number analyzed (Participants) | 69 | 43
m/sec | 0.9 (0.24) | 0.9 (0.17)
Statistical Analysis 1: Comparison: Population: II BYM338 700 mg vs Population: II Placebo; Population II: Gait speed at Week 49; Test type: Other; p = 0.395, ANCOVA; Difference in the least square means (SE)

7. Secondary Outcome: Population I: Appendicular Skeletal Muscle Index (ASMI) as Measured by Dual Energy X-ray Absorptiometry (DXA) at Week 49
Description: ASMI is a core requirement for determining the presence of sarcopenia and is calculated as the sum of the appendicular lean mass (kg) of the two upper and two lower limbs quantified by DXA, divided by height (m2). Therefore, an increase in ASMI indicates an increase in the quantity of an individual's lean mass.
Time Frame: Week 49
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg/m^2
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15
kg/m^2 | 6.6 (7.22) | 6.0 (14.05) | 6.1 (8.08) | 5.8 (15.08) | 5.9 (14.19) | 5.2 (14.85) | 5.6 (15.21)
Statistical Analysis 1: Comparison: Population I: BYM338 700 mg vs Population I BYM338: 700 mg to Placebo; Population I: ASMI at Week 49; Test type: Other; p = 0.120, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 2: Comparison: Population I: BYM338 210 mg vs Population I BYM338: 210 mg to Placebo; Population I: ASMI at Week 49; Test type: Other; p = 0.297, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 3: Comparison: Population I: BYM338 70 mg vs Population I: BYM338 70 mg to Placebo; Population I: ASMI at Week 49; Test type: Other; p = 0.074, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 4: Comparison: Population I: BYM338 700 mg vs Population I: Placebo; Population I: ASMI at Week 49; Test type: Other; p = 0.022, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 5: Comparison: Population I: BYM338 210 mg vs Population I: Placebo; Population I: ASMI at Week 49; Test type: Other; p = 0.106, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 6: Comparison: Population I: BYM338 70 mg vs Population I: Placebo; Population I: ASMI at Week 49; Test type: Other; p = 0.211, t-test, 1 sided; One-sided test at the 0.025 significance level

8. Secondary Outcome: Population II: Appendicular Skeletal Muscle Index (ASMI) as Measured by Dual Energy X-ray Absorptiometry (DXA) at Week 49
Description: as for outcome 7
Time Frame: Week 49
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg/m^2
Arm/Group | Population: II BYM338 700 mg | Population: II Placebo
Number analyzed (Participants) | 69 | 43
kg/m^2 | 5.6 (14.36) | 5.5 (12.46)
Statistical Analysis 1: Comparison: Population: II BYM338 700 mg vs Population: II Placebo; Population II: ASMI at Week 49; Test type: Other; p = 1.000, ANCOVA; Difference in the least square geometric means

9. Secondary Outcome: Population I: Total Lean Body Mass (LBM) as Measured by Dual Energy X-ray Absorptiometry (DXA) at Week 49
Description: LBM is defined as the Total soft tissue fat-free body mass. A high LBM represents better pharmacodynamic effect
Time Frame: Week 49
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg
Arm/Group | Population I: BYM338 700 mg | Population I BYM338: 700 mg to Placebo | Population I: BYM338 210 mg | Population I BYM338: 210 mg to Placebo | Population I: BYM338 70 mg | Population I: BYM338 70 mg to Placebo | Population I: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 7 | 15
kg | 41.4 (21.11) | 34.0 (17.76) | 35.5 (15.39) | 32.6 (25.23) | 34.9 (21.16) | 34.0 (18.47) | 32.6 (17.95)
Statistical Analysis 1: Comparison: Population I: BYM338 700 mg vs Population I BYM338: 700 mg to Placebo; Population I: LBM at Week 49; Test type: Other; p = 0.084, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 2: Comparison: Population I: BYM338 210 mg vs Population I BYM338: 210 mg to Placebo; Population I: LBM at Week 49; Test type: Other; p = 0.283, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 3: Comparison: Population I: BYM338 70 mg vs Population I: BYM338 70 mg to Placebo; Population I: LBM at Week 49; Test type: Other; p = 0.323, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 4: Comparison: Population I: BYM338 700 mg vs Population I: Placebo; Population I: LBM at Week 49; Test type: Other; p = 0.018, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 5: Comparison: Population I: BYM338 210 mg vs Population I: Placebo; Population I: LBM at Week 49; Test type: Other; p = 0.179, t-test, 1 sided; One-sided test at the 0.025 significance level
Statistical Analysis 6: Comparison: Population I: BYM338 70 mg vs Population I: Placebo; Population I: LBM at Week 49; Test type: Other; p = 0.227, t-test, 1 sided; One-sided test at the 0.025 significance level

10. Secondary Outcome: Population II: Total Lean Body Mass (LBM) as Measured by Dual Energy X-ray Absorptiometry (DXA) at Week 49
Description: LBM is defined as the Total soft tissue fat-free body mass. A high LBM represents better pharmacodynamic effect
Time Frame: Week 49
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg
Arm/Group | Population: II BYM338 700 mg | Population: II Placebo
Number analyzed (Participants) | 69 | 43
kg | 34.9 (25.01) | 33.7 (20.40)
Statistical Analysis 1: Comparison: Population: II BYM338 700 mg vs Population: II Placebo; Population II: LBM at Week 49; Test type: Other; p = 1.000, ANCOVA; Difference in the least square geometric means

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum treatment duration of 24 weeks
Description: Adverse events presented below are events considered to be treatment-emergent, therefore only events occurring in Population I are summarized. Patients in Population II did not receive study medication (were followed-up of-drug), thus any events occurring in this group were not treatment-emergent and are not captured in the summary.
Groups:
- Population I BYM338 700 mg; Population I BYM338 700 mg to Placebo; Population I BYM338 210 mg; Population I BYM338 210 mg to Placebo; Population I BYM338 70 mg; Population I BYM338 70 mg to Placebo; Population I Placebo: Follow-up (arm 1): Patients in Population I received 6 doses of bimagrumab 70 mg, 210 mg, 700 mg or placebo - one approximately every four weeks - over a 20-week period providing drug exposure for a total of 24 weeks.
Arm/Group | Population I BYM338 700 mg | Population I BYM338 700 mg to Placebo | Population I BYM338 210 mg | Population I BYM338 210 mg to Placebo | Population I BYM338 70 mg | Population I BYM338 70 mg to Placebo | Population I Placebo | Population: II BYM338 700 mg | Population: II Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/7 | 0/7 | 0/15 | 0/69 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/5 | 0/4 | 0/7 | 2/7 | 2/15 | 0/69 | 0/43
Other Adverse Events (participants affected / at risk) | 4/5 | 4/5 | 3/5 | 2/4 | 5/7 | 3/7 | 11/15 | 0/69 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Population I BYM338 700 mg (N=5) | Population I BYM338 700 mg to Placebo (N=5) | Population I BYM338 210 mg (N=5) | Population I BYM338 210 mg to Placebo (N=4) | Population I BYM338 70 mg (N=7) | Population I BYM338 70 mg to Placebo (N=7) | Population I Placebo (N=15) | Population: II BYM338 700 mg (N=69) | Population: II Placebo (N=43)
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Population I BYM338 700 mg (N=5) | Population I BYM338 700 mg to Placebo (N=5) | Population I BYM338 210 mg (N=5) | Population I BYM338 210 mg to Placebo (N=4) | Population I BYM338 70 mg (N=7) | Population I BYM338 70 mg to Placebo (N=7) | Population I Placebo (N=15) | Population: II BYM338 700 mg (N=69) | Population: II Placebo (N=43)
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2 | 0 | 6 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body mass index decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device loosening (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02468674/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT02468674/SAP_001.pdf